CLINICAL TRIAL: NCT02051673
Title: Induction of Donor-Specific Tolerance in Recipients of Live Donor Stem Cell Infusion (Compassionate Use)
Status: No longer available | Type: Expanded Access
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: ICT-7392-Compassionate Use
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Renal Failure
Keywords: Kidney Transplantation
MeSH Terms: conditions — Renal Insufficiency | interventions — Biological Products

INTERVENTIONS:
Biological: Biological/Vaccine: Enriched Hematopoetic Stem Cell Infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
Four subjects were treated under compassionate use provisions under this study with facilitating cell therapy (FCRx)

DETAILED DESCRIPTION:
Four subjects were treated under compassionate use provisions under this study with facilitating cell therapy (FCRx) and living donor kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between the ages of 18 and 65 years and meet the institution's criteria for renal transplantation for end-organ failure
* Patient is receiving first renal transplant
* Patient is receiving a renal transplant only
* The crossmatch is negative between donor and recipient
* Women who are of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours of initiating total body irradiation (TBI) and agree to use reliable contraception for 1 year following transplant
* Potential donors who are women of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours prior to receiving Granulocyte colony-stimulating factor (G-CSF)
* No evidence of donor-specific antibody presently or historically

Exclusion Criteria:

* Clinically active bacterial, fungal, viral or parasitic infection
* Pregnancy
* Clinical or serologic evidence of viral infection which would preclude the recipient from receiving a kidney transplant
* Previous radiation therapy at a dose which would preclude TBI
* Positive crossmatch between donor and recipient
* Evidence for immunologic memory against donor
* BMI >35 or <18
* Re-transplant
* Positive serologies for hepatitis B virus (HBV), hepatitis C virus (HCV), HIV

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States